CLINICAL TRIAL: NCT01361815
Title: A Prospective Multicenter Trial to Explore the Tolerability and Safety of the H-Coil Deep TMS in Combination With Serotonin Selective Reuptake Inhibitor(SSRI) for Subjects With MDD Who Complete/ Discontinued the CTP-0001-00 Protocol
Brief Title: Prospective Multicenter Trial to Explore the Tolerability and Safety of the H-Coil Deep TMS in Combination With Serotonin Selective Reuptake Inhibitor(SSRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-0002-00
Record Dates: First submitted 2011-05-26; First posted 2011-05-27 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2015-02

CONDITIONS: Major Depressive Disorder, Recurrent, Unspecified; Major Depressive Disorder, Single Episode, Unspecified
Keywords: Depression; MDD; SSRIs; TMS
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- H-Coil Deep TMS Treatment (Other)
  Interventions: Device: H-Coil Deep TMS in combination with SSRIs

INTERVENTIONS:
Device: H-Coil Deep TMS in combination with SSRIs — The study group will receive DTMS treatment three times a week for four weeks in combination with SSRI medications.
  Other Names: H-Coil Deep TMS Treatment

SUMMARY:
The purpose of the study is to explore the Tolerability and Safety of the H-Coil deep Transcranial Magnetic Stimulation (TMS) in combination with Serotonin Selective Reuptake Inhibitor (SSRI) for Subjects with Major Depression Disorder (MDD) who Complete/ Discontinued the Deep TMS Multicenter study for Subjects with Major Depression Disorder (MDD) (Protocol# CTP-0001-00).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Men and women 22-68 years of age
* Primary DSM-IV diagnosis of Major Depression, single or recurrent episode confirmed by the Structured Clinical Interview for the DSM-IV (SCID-IV).
* Completed the CTP-0001-00 study according to the protocol, i.e., either completed 16 weeks of treatment, or were discontinued from the CTP-0001-00 study protocol after 6 weeks or more from randomization.
* Capable and willing to provide informed consent.
* Able to adhere to the treatment schedule.

Exclusion Criteria:

* Discontinued from CTP-0001-00 study protocol due to the following reasons: Tolerability and safety reason, Non-compliant with the study protocol, Developed documented suicidal ideation as assessed by the investigator or significant suicide risk based on HDRS-21 item 3 score of 3 or 4 or suicidal attempt
* Current psychotic disorder
* Sensitivity or allergic or other severe adverse event previously reported for Citalopram, Escitalopram, Fluoxetine, Paroxetine, or Sertraline.
* Known or suspected pregnancy
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.
* Minimal MT found for both hands is higher than 75% of stimulator power output.

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The tolerability and safety of H-coil deep rTMS treatment in combination with SSRI medications | 4 weeks
  Safety:
  AE incidence, Vital signs, Physical and neurological examination, Young Manic Rating Scale (YMRS), Suicide Ideation Scale (SSI)
  Tolerability:
  Number of subjects (%) who discontinue the study, Number of subjects (%) who discontinue the study due to AEs

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Zangan, Prof., Principal Investigator — Weizmann Institute of Science; Yechiel Levkovitz, Prof., Principal Investigator — Shalvata Mental Health Center
Locations (19):
- United States (13):
  - UC Davis Center for Mind & Brain, Davis, California
  - University of California (UCLA), Los Angeles, California
  - Smart Brain and Health, Santa Monica, California
  - Advanced Mental Health Care Inc. - Juno Beach, Juno Beach, Florida
  - Advanced Mental Health Care Inc. - Royal Palm Beach, Royal Palm Beach, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - McLean Hospital - TMS Services, Belmont, Massachusetts
  - Greater Nashua Mental Health Center, Nashua, New Hampshire
  - Neuropharmacology Services, New York, New York
  - Columbia University / New York State Psychiatric Institute, New York, New York
  - Medical Uni. Of South Carolina (MUSC), Charleston, South Carolina
  - Senior Adults Specialty Research, Austin, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
- Center for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada
- Germany (2):
  - Universitätsklinikum Bonn, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Bonn
  - Klinik für Psychiatrie und Psychotherapie, Ludwig-Maximilians-Universität, Munich
- Israel (3):
  - Beer Yaacov Mental Health Center, Be’er Ya‘aqov
  - Shalvata Mental Health Center, Hod HaSharon
  - Hadasah Ein-Karem Medical Center, Jerusalem